CLINICAL TRIAL: NCT03056664
Title: The Safety and Efficiacy of Local MSC Injection in the Treatment of Fistulas in Patients With Perianal Crohn's Disease
Brief Title: The Role of MSC in the Treatment of Fistulas in Patients With Perianal Crohn's Disease
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MSCINCDGL
Record Dates: First submitted 2015-08-24; First posted 2017-02-17 (Actual); Last update posted 2017-02-17 (Actual); Status verified 2016-09

CONDITIONS: Crohn's Disease; Fistula
MeSH Terms: conditions — Crohn Disease; Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- MSC-1 (Experimental): Patient in this arm will receive routine surgery and local MSC injection of 3×10E6/kg
  Interventions: Procedure: Routine drainage surgery; Biological: MSC injection 01
- MSC-2 (Experimental): Patient in this arm will receive routine surgery and local MSC injection of 6×10E6/kg
  Interventions: Procedure: Routine drainage surgery; Biological: MSC injection 02
- Ctrl (Experimental): Patient in this arm will receive routine surgery and local NS injection
  Interventions: Procedure: Routine drainage surgery; Other: placebo

INTERVENTIONS:
Procedure: Routine drainage surgery
Biological: MSC injection 01 — Local MSC injection in peri-anal with a dose of 3×10E6/kg
  Arms: MSC-1
Biological: MSC injection 02 — Local MSC injection in peri-anal with a dose of 6×10E6/kg
  Arms: MSC-2
Other: placebo — NS injection instead of MSC
  Arms: Ctrl

SUMMARY:
Here investigators will carry out this phase II clinical trial to explore a effective therapeutic regimen of MSC in the Crohn's perianal fistula.

DETAILED DESCRIPTION:
Peri-anal fistula is common seen in Crohn's disease. Treatments including surgery, antibiotics, immunosuppressive drug and infliximab improve the quality of life of the patients suffering Crohn's perianal fistula, but the recurrent rate is still high. MSC showed promising effect in the therapy of CD, but the standard treatment strategy is unclear. Here investigators will carry out this phase II clinical trial to explore a effective therapeutic regimen of MSC in the Crohn's perianal fistula.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years old, male or female;
2. refractory CD fistula, there are 1-2 and 1-3 in the mouth fistula;
3. Diagnostic CD at least three months;
4. CDAI <250;
5. were receiving drug treatment (5-ASA and hormones> 4 weeks, immunosuppressants and biological agents> 8 weeks);
6. signed informed consent.

Exclusion Criteria:

1. with intestinal obstruction, stenosis, or perianal abscess;
2. pregnant or lactating women;
3. infection needs antibiotics persons;
4. rectovaginal fistula;
5. complex anal fistula more than two inside the mouth;
6. stenosis or perforation CD;
7. perianal infection;
8. could not do rectal or anal stenosis local injection therapy;
9. with acute enteritis;
10. , liver and kidney dysfunction;
11. a month have used other drugs are in clinical trials;
12. no conditions or unwilling to carry out MRI inspected;
13. who are adjusting therapy;
14. HIV patients;
15. The combined active hepatitis or tuberculosis; Occurred in 16) 6 months opportunistic infections, or severe infections occur within three months;

17) In the past five years, those who suffer from cancer; 18) there is a history of lymphoproliferative disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2017-01; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Clinical response(fistula closure) | 12 weeks
  Physical examination indicates fistula healing, or MRI examinations showed fistula healing more than 2cm

SECONDARY OUTCOMES:
C-reactive protein (CRP) | 12 weeks
  To summarize the changes from baseline compared to 12 weeks in serum C-reactive protein (CRP)
Clinical Response | 6 weeks after receiving treatment
  CDAI means Crohn's Disease Activity Index.The purpose of this crohn's disease activity index (CDAI) calculator is to gauge the progress or lack of progress for people with crohn's disease. The reference article says "generally speaking, CDAI scores below 150 indicate a better prognosis than higher scores." Clinical Response of patients 6 weeks after receiving treatment (CDAI score less than 150)